CLINICAL TRIAL: NCT03659188
Title: Evaluation of the Efficiency and Efficacy of Flapless Cortico-alveolar Perforations Using Mechanical Drills Versus Traditional Corticotomy in the Retraction of Upper Canines: a Three-arm Randomized Controlled Clinical Trial
Brief Title: Comparison Between Two Methods in the Acceleration of the Retraction of Upper Canines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-18-2018
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Malocclusion, Angle Class II, Division 1
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cortico-alveolar perforations (Experimental): Patients will undergo orthodontic treatment plus cortico-alveolar perforations.
  Interventions: Procedure: Cortico-alveolar perforations
- Traditional Corticotomy (Experimental): Patients will undergo orthodontic treatment plus an acceleration procedure employing traditional corticotomy.
  Interventions: Procedure: Traditional Corticotomy
- Control (No Intervention): Patients will undergo orthodontic treatment in which canine retraction will be accomplished using the standard sliding mechanism without any acceleration procedures.

INTERVENTIONS:
Procedure: Cortico-alveolar perforations — Mechanical drills will be used on a handpiece
  Other Names: Flapless corticotomy
  Arms: Cortico-alveolar perforations
Procedure: Traditional Corticotomy — Piezo-surgery will be employed following flaps' elevation.
  Arms: Traditional Corticotomy

SUMMARY:
Patients at the Orthodontic Department of University of Damascus Dental School will be examined and subjects who meet the inclusion criteria will be included.

Then, initial diagnostic records (diagnostic gypsum models, internal and external oral photographs, as well as radiographic images) will be studied to ensure that the selection criteria are accurately matched.

The aim of this study is to compare flapless bone cutting by mechanical drills to evaluate the acceleration of the retraction of upper canines versus traditional bone cutting by piezo-surgery in comparison with a control group without bone cutting after extraction of upper first premolars in class II type I patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-27 years
* Patients who have malocclusion class II type I and who require first-premolar extraction with:
* Dentoalveolar class II type I with ANB between 5 and 9 degrees.
* Protrusion between (5-10 mm)
* Overbite between (0-4)
* Vertical dimension is normal or over the normal range
* Mild to moderate crowding
* All patients should have complete permanent occlusion on the maxilla
* All patients should have normal periodontal tissue and good oral health, which will be assessed by:

  1. Depth of the gingival pocket does not exceed 4 mm
  2. Plaque index does not exceed 1
  3. Gingival index does not exceed 1

Exclusion Criteria:

* Patients in which oral surgery under local anesthesia is contraindicated due to medical, psychological, or social reasons.
* Patients who have a general health problem that affects dental movement
* Patients who have undergone previous orthodontic treatment
* Patients with mixed occlusion
* Patients who have lost one or more of their teeth since birth or who have one of the permanent teeth extracted (except the third molar)
* Patients who have bad oral health or active periodontal disease

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Change in Canine Retraction Speed | T1: At the end of alignment (which is expected within 3 months); T2: 1 month after canine retraction; T3: After two months; T4: After 3 months; T5: at the end of canine retraction which is expected within 5 months
  The rate at which canine is going to be retracted (mm/month) in each group will be calculated.
  This outcome will be measured by the following steps:
  1. Drawing a projection from the upper canine apex to the middle palatal bone line.
  2. Drawing a projection from the mesial ending of the third palatal rugae to the middle palatal bone line.
  3. Measuring the distance (mm) between the two orthogonal projections.
  4. The rate of canine retraction will be measured by dividing the distance between the two orthogonal projections by the time elapsed between assessment times.
Change in Anchorage Loss | T1: At the end of alignment (which is expected within 3 months); T2: 1 month after canine retraction; T3: After two months; T4: After 3 months; T5: at the end of canine retraction which is expected within 5 months
  Anchorage loss in related the mesial drift of the first molar. This outcome will be measured by drawing two projections from the central groove of the first maxillary molar and the mesial ending of the third palatal rugae to the middle palatal bone line. The mesial migration of the first maxillary molar (mm) will be measured by dividing the distance between the two projections by the time elapsed between assessment times.
Change in Canine Rotation | T1: At the end of alignment (which is expected within 3 months); T2: 1 month after canine retraction; T3: After two months; T4: After 3 months; T5: at the end of canine retraction which is expected within 5 months
  The angle between the middle palatal bone and the line through the mesial and distal edges of the canine will be measured on each side. The rotation will be assessed by calculating the difference between the angles on two different times. Then, the speed of rotation will be calculated by dividing the rotation angle (degrees) by time that elapsed between assessment times.
Change in Canine Axis | T1: at the end of the alignment stage (which is expected within 3 to 4 months); T2: at the end of the canine retraction stage (which is expected to occur with 4 to five months following the onset of this stage).
  The changes in the canine axis during retraction will be studied by calculating canine angulation (arithmetic mean of the angulation of the right and left upper canine axis with the anterior cranial base plane) on lateral cephalometric radiographs. The difference between the canine angulation on T1 and T2 will be calculated after comparing the two cephalometric using Viewbox version 4.0.0.98.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Al-Bitar, DDS MSc, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental School, Damascus, Syria; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Bassel Brad, DDS MSc PhD, Study Director — Associate Professor of Oral and Maxillofacial Surgery, Oral and Maxillofacial Surgery Department, University of Damascus Dental School, Damascus, SYRIA
Locations (1):
- Orthodontic Department, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbas NH, Sabet NE, Hassan IT. Evaluation of corticotomy-facilitated orthodontics and piezocision in rapid canine retraction. Am J Orthod Dentofacial Orthop. 2016 Apr;149(4):473-80. doi: 10.1016/j.ajodo.2015.09.029. PMID 27021451
- [Background] Alfawal AM, Hajeer MY, Ajaj MA, Hamadah O, Brad B. Effectiveness of minimally invasive surgical procedures in the acceleration of tooth movement: a systematic review and meta-analysis. Prog Orthod. 2016 Dec;17(1):33. doi: 10.1186/s40510-016-0146-9. Epub 2016 Oct 24. PMID 27696311
- [Background] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579
- [Background] Aksakalli S, Calik B, Kara B, Ezirganli S. Accelerated tooth movement with piezocision and its periodontal-transversal effects in patients with Class II malocclusion. Angle Orthod. 2016 Jan;86(1):59-65. doi: 10.2319/012215-49.1. Epub 2015 May 19. PMID 25989211
- [Background] Buyuk SK, Yavuz MC, Genc E, Sunar O. A novel method to accelerate orthodontic tooth movement. Saudi Med J. 2018 Feb;39(2):203-208. doi: 10.15537/smj.2018.2.21235. PMID 29436571